CLINICAL TRIAL: NCT02095821
Title: Observational Study of Fibrinogen as a Surrogate for Global Haemostasis in Plasma Exchange Therapy
Brief Title: Fibrinogen as a Surrogate for Global Haemostasis in Plasma Exchange
Status: Terminated | Type: Observational
Why Stopped: Study was stopped due to recruitment failure
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Julius Schmidt, MD, Hannover Medical School
Other Study IDs: FIB-2110-2014
Record Dates: First submitted 2014-02-27; First posted 2014-03-26 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Clotting Disorder Due to Plasma Exchange Therapy; Humoral Rejection After Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Humoral rejection, TPE

SUMMARY:
Plasma exchange is a frequently used therapy in many antibody-mediated disorders, such as humoral rejection after kidney transplantation. Treatment frequency is adjusted to daily measured fibrinogen blood levels to prevent bleeding complications. However, data about the correlation of fibrinogen blood levels and function of the coagulation system during plasma exchange therapy is scarce. In the present study we examine blood fibrinogen levels and coagulation factors as well as thrombin clotting time in patients under plasma exchange therapy.

ELIGIBILITY:
Inclusion Criteria:

* plasma exchange therapy due to humoral rejection after kidney transplantation

Exclusion Criteria:

* hereditary coagulopathy
* chronic liver disease (Child C)
* therapeutic anticoagulation
* malnutrition (BMI<17.5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary hospital patients after kidney transplantation, humoral rejection
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Thrombin clotting time | Baseline, daily measurement until hospital discharge (avarage hospital stay: 10 days)
  Daily measurement after initiation of plasma exchange therapy until treatment course is finished

CONTACTS AND LOCATIONS:
Overall Officials: Sascha David, MD, Principal Investigator — Medical School Hannover
Locations (1):
- Hannover Medical School, Hanover, Germany